CLINICAL TRIAL: NCT00151528
Title: A Long-Term, Open-Label, Safety Trial of Pregabalin in Patients With Fibromyalgia
Brief Title: An Open-Label Trial of Pregabalin in Patients With Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081057
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2006-07

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
The main purpose of this protocol is to evaluate the long-term safety of pregabalin in patients who participated in the previous fibromyalgia Study A0081056 and who wish to receive open-label pregabalin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met the inclusion criteria for the preceding fibromyalgia Protocol A0081056
* Must have received pregabalin/placebo under double-blind conditions.

Exclusion Criteria:

* Patients may not participate in the study if they experienced a serious adverse event during the previous fibromyalgia Study A0081056 which was determined to be related to the study medication by the investigator or the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428
Dates: Start 2005-01; Study Completion 2006-06

PRIMARY OUTCOMES:
Main outcome of the study is long-term safety of pregabalin in patients with fibromyalgia. This is a 1 year open-label extension of the preceding double-blind randomized fibromyalgia protocol A0081056.

SECONDARY OUTCOMES:
There are no secondary outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (81):
- United States (81):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Los Alamitos, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Pismo Beach, California
  - Pfizer Investigational Site, Redondo Beach, California
  - Pfizer Investigational Site, Riverside, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Whittier, California
  - Pfizer Investigational Site, Danbury, Connecticut
  - Pfizer Investigational Site, New Milford, Connecticut
  - Pfizer Investigational Site, Stratford, Connecticut
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Palm Beach Gardens, Florida
  - Pfizer Investigational Site, Seminole, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Sunrise, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Maywood, Illinois
  - Pfizer Investigational Site, Oak Brook, Illinois
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Newton, Massachusetts
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Lansing, Michigan
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Princeton, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Wilmington, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Mogadore, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Johnstown, Pennsylvania
  - Pfizer Investigational Site, Mechanicsburg, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Pottstown, Pennsylvania
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, Wyomissing, Pennsylvania
  - Pfizer Investigational Site, Anderson, South Carolina
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Lubbock, Texas
  - Pfizer Investigational Site, Richardson, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Woodstock, Vermont
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Yakima, Washington

REFERENCES:
- [Derived] Arnold LM, Emir B, Murphy TK, Zeiher BG, Pauer L, Scott G, Petersel D. Safety profile and tolerability of up to 1 year of pregabalin treatment in 3 open-label extension studies in patients with fibromyalgia. Clin Ther. 2012 May;34(5):1092-102. doi: 10.1016/j.clinthera.2012.03.003. Epub 2012 Apr 14. PMID 22503162
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081057&StudyName=An+Open%2DLabel+Trial+of+Pregabalin+in+Patients+with+Fibromyalgia+++